CLINICAL TRIAL: NCT04715412
Title: Impact of Clinical Pharmacy Guided Patient Counseling and Adherence Support on Renal Transplant Recipients' Adherence and Health Outcomes
Brief Title: Clinical Pharmacy Guided Patient Counselling and Adherence Support on Renal Transplant Recipients
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Future University in Egypt (Other)
Collaborators: Ain Shams University (Other)
Responsible Party: Principal Investigator, Doaa Mohamed Salah ElDin Diab ELBohy, Assistant professor of Clinical Phramcy, Future University in Egypt
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Health Services Research
Other Study IDs: REC-ASU No 10
Record Dates: First submitted 2021-01-14; First posted 2021-01-20 (Actual); Last update posted 2021-01-20 (Actual); Status verified 2021-01

CONDITIONS: Transplant;Failure,Kidney

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Study group (Other): The standard training sessions were conducted for individual patient by the transplant physician to explain rejections, infections and tumor risks, post-transplant medication. After discharge, all patients had scheduled follow-up visits at the outpatient clinic of the transplant center, where immune suppressant blood levels were measured and their dosing adjusted accordingly. Patients also had the opportunity to discuss any concern of their condition or drug therapy with the transplant physician in charge.
  in addition to this standard transplant training, patients received intensified care by a dedicated clinical pharmacist combining educational and technical interventions aiming at achieving and maintaining adherence to his/her prescribed medication and improving health outcomes.
  Interventions: Other: patient counseling and adherence support

INTERVENTIONS:
Other: patient counseling and adherence support — Technical interventions include; identification of possible reasons for non-adherence, adherence support by developing simplified schedules for taking medications that were customized to individualized patient's lifestyle. Reminders for dose as well as tools/strategies the RTR may use to follow the dosing schedules if needed as pillbox were provided as needed
  Clinical pharmacists' guided patient training was individualized, repetitive, covered 6 months, and included more aspects and provided practical hints and strategies for medication management.
  Initial clinical pharmacist face-to-face session will be up to 60-minute then 30-minute follow-up sessions will be conducted monthly for 6 months during the scheduled post-transplant clinic visits as coordinated with the transplant physician to allow for single office visits for transplant related issues and comorbidities.

SUMMARY:
As a result of the shortage of donor organs and the close relationship between allograft or even life loss and non-adherence after kidney transplantation, improvement of patient adherence appears essential. So the current study aimed to monitor adherence barriers of renal transplant recipients and evaluate possible consequences of nonadherence on recipients' clinical outcomes as well as to implement a structured adherence management program consisting of intensified patient counselling and adherence support by a dedicated clinical pharmacist as an adjunct to standard post-transplant patient education carried out by transplant physicians to investigate the efficacy of the implemented program on patients adherence and health outcomes as compared to standard physician patient care. The study is a prospective self-controlled interventional study that recruited 69 living donors-renal transplant Patients attending the transplant clinic of Nasser institute and satisfying the inclusion criteria. On enrolment, patient-related baseline data that could determine and affect patients' adherence as well as patients' clinical outcomes were recorded. After all patients received the adjuvant adherence management program by the clinical pharmacist for 6 month, patients' health outcomes were re-evaluated to compare them to baseline data

ELIGIBILITY:
Inclusion Criteria:

>18 years at least 1 year post-transplant to allow for stabilization of the prescribed immunosuppressant therapy (IST) regimen Independent of others for medication management and willing as well as able to repetitively visit the outpatient clinic for educational training & data collection.

Exclusion Criteria:

* Pediatric Older than 65 years. Multi-organ transplant. Pregnant or lactating. Cancer patients.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2020-03-10 (Actual); Primary Completion 2020-11-11 (Actual); Study Completion 2020-12-31 (Actual)

PRIMARY OUTCOMES:
Specified clinical and educational outcome | 6 months
  Self-reported taking adherence [TA, percentage of doses taken in comparison to the total number of doses prescribed]. Patients will be classified as being adherent for those with TA ≥80 or non-adherent for those with TA <80

SECONDARY OUTCOMES:
Renal function | 6 months
  Serum creatinine mg/dL
Renal function | 6 months
  BUN (blood urea nitrogen) mg/dL
Renal function | 6 months
  Serum uric acid mg/dL Serum uric acid
Serum trough Immunosuppressant level (C0) | 6 months
  Serum level of immunosuppressant
CBC | 6 months
  blood sample to asses (RBCs, WBCs and platelets)

CONTACTS AND LOCATIONS:
Locations (1):
- Transplantation Clinic Nasser Institute, Cairo, Egypt

IPD SHARING:
Plan to Share IPD: No